CLINICAL TRIAL: NCT04715152
Title: Adductor Canal Block Versus Intra-articular Analgesia for Postoperative Pain After Arthroscopic Anterior Cruciate Ligament Reconstruction: a Randomized Trial
Brief Title: ACB Versus IA Analgesia in Knee Arthroscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Seham Mohamed Moeen Ibrahim, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SM 1 2021
Record Dates: First submitted 2021-01-15; First posted 2021-01-20 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACB group (Active Comparator): Patients will receive ultrasound-guided (USG) ACB with bupivacaine and dexamethasone 30 minutes before spinal anesthesia and sham intra-articular normal saline.
  Interventions: Drug: ACB group
- IA group (Placebo Comparator): Patients will receive intra-articular bupivacaine and dexamethasone at the end of surgery and sham USG-ACB with normal saline.
  Interventions: Drug: IA group

INTERVENTIONS:
Drug: ACB group — Patients will receive ultrasound-guided (USG) ACB with bupivacaine and dexamethasone 30 minutes before spinal anesthesia and sham intra-articular normal saline
  Arms: ACB group
Drug: IA group — Patients will receive intra-articular bupivacaine and dexamethasone at the end of surgery and sham USG-ACB with normal saline
  Arms: IA group

SUMMARY:
Reconstruction of the anterior cruciate ligament (ACL) of the knee is a painful procedure, and effective postoperative analgesia is important for early return of patient activity.

DETAILED DESCRIPTION:
Reconstruction of the anterior cruciate ligament (ACL) of the knee is a painful procedure, with postoperative analgesia providing patient comfort, early mobilization, and discharge within 24 hours.

Various methods for postoperative analgesia management are available, such as systemic opioids, epidural local anesthetic, peripheral nerve block and local anesthetic infiltration analgesia. Use of systemic opioids can cause adverse effects that may affect functional rehabilitation, such as nausea, vomiting, pruritus, sedation and respiratory depression. Hypotension, urinary retention, and pruritus are more common in patients with epidural analgesia. In addition, use of long-acting intrathecal opioids causes adverse effects such as bilateral motor block, tremor and hypotension. Systemic and intrathecal methods for postoperative analgesia are gradually being abandoned because of these negative effects.

The saphenous nerve is the largest contributor to sensory perception around the knee, while the adductor canal contains the nerve to the vastus medialis, the medial femoral cutaneous nerve, the medial retinacular nerve, articular branches from the posterior division of the obturator nerve and occasionally the anterior branch of the obturator nerve. Although adductor canal block (ACB) can contribute towards motor blockade of the periarticular musculature, its effect on functional weakness of the quadriceps has been reported to be minimal, compared with femoral nerve block (FNB).

Intra-articular (IA) local anesthetic agents have been used either alone or in combination with other agent. However, it was observed that use of combination of drug is better than single drug for prevention of postoperative pain, providing synergistic effect and reducing side effects compared to high dose of single drug.

Dexamethasone is a potent and highly selective glucocorticoid with minimal mineralocorticoid effect. It blocks the nociceptive impulse transmission along the myelinated C fibers. Dexamethasone prolongs the duration of regional blocks, when combined with local anesthetics.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective arthroscopic reconstruction of the anterior cruciate ligament (ACL) under spinal anesthesia, aged from 18 to 65 years old

Exclusion Criteria:

* Contraindications to peripheral nerve block (e.g. allergy to local anesthetics, coagulopathy, infection in the area)
* History of cardiovascular, cerebrovascular, and respiratory diseases
* Preexisting neuropathies
* Chronic pain syndrome
* Opioid dependence
* Patients with diabetes mellitus, sever hypertension, hepatic or renal dysfunction
* Pregnancy
* Not willingness to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
The pain free time after surgery | 1440 minutes (24 hours) after surgery
  assessed in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Seham M Moeen, MD, Principal Investigator — Assiut University
Locations (1):
- Seham Mohamed Moeen, Asyut, Egypt